CLINICAL TRIAL: NCT03124186
Title: Sensory-driven Motor Recovery in Poorly Recovered Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumy Sawaki (Other)
Responsible Party: Sponsor-Investigator, Lumy Sawaki, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5R01HD056002 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: motor recovery; neuroplasticity; subacute; human; sensory; nerve stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation with motor training (Experimental): 2 hours of active peripheral nerve stimulation (intervention) paired with 4 hours of intensive task-oriented upper extremity training. Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy. Peripheral nerve stimulation will be delivered using a S88 Dual Output Stimulator by Grass Technologies.
  Interventions: Device: S88 Dual Output Stimulator by Grass Technologies
- Sham stimulation with motor training (Active Comparator): 2 hours of sham peripheral nerve stimulation (intervention) paired with 4 hours of intensive task-oriented upper extremity training. Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy. Peripheral nerve stimulation will be delivered using a S88 Dual Output Stimulator by Grass Technologies.
  Interventions: Device: S88 Dual Output Stimulator by Grass Technologies

INTERVENTIONS:
Device: S88 Dual Output Stimulator by Grass Technologies — Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy

SUMMARY:
This research project addresses a scientifically important question that cannot be answered by other means. The use of peripheral nerve stimulation has the potential to enhance recovery in subacute stroke patients with poor functional recovery. The primary objective of this proposal is to demonstrate that peripheral nerve stimulation combined with intensive motor training has the ability to further improve hand motor function when compared to intensive training alone or nerve stimulation alone. The results from this study have the potential to develop new strategies in neurorehabilitation.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability in the United States. Approximately 70-88% of persons with ischemic stroke have some degree of motor impairment. A major goal of research in stroke rehabilitation is to harness the ability of the brain to reorganize after neurologic damage has occurred and thus ultimately lead to successful recovery of function. Data from animal and human models have suggested that sensory input plays an important role in motor output, possibly by influencing cortical plasticity. However, in spite of the advances to date, little is known about the extent to which sensory input in the form of peripheral nerve stimulation (PNS) can be successfully combined to physical training, especially in poorly recovered subacute stroke patients. The proposed study will evaluate the effectiveness of sustained PNS coupled with motor training, to improve hand motor function in subacute stroke patients with severe motor deficit. Our preliminary data in chronic stroke patients with severe motor deficit demonstrate that motor function can be substantially enhanced when PNS is paired with motor training. In addition, a separate study in patients with mild motor deficit receiving motor training alone suggests that the optimal therapeutic time window to deliver motor training is within the first year after stroke. The improvement of behavioral motor function was associated with corticomotor reorganization. Therefore, this study proposes to evaluate the effectiveness of sustained PNS paired with motor training, to promote functional motor recovery in subacute stroke patients with severe motor deficit. The central hypothesis is that subacute stroke patients with severe motor deficit receiving PNS and intensive task-oriented therapy will have improved motor function compared to patients receiving sham-PNS and task-oriented therapy, and the degree of this behaviorally-measured effect will correlate with the neurophysiological effect measured by transcranial magnetic stimulation. The investigators plan to accept or reject the central hypothesis by accomplishing two Specific Aims: 1) test the effect of PNS preceding task-oriented therapy on hand motor function, and 2) test the effect of PNS preceding task-oriented therapy on motor map measured by transcranial magnetic stimulation. The long-range goals are: a) to maximize the restoration of hand motor function after stroke, b) to determine the impact of this intervention in activities of daily living, and c) collect solid data to prepare for a future multicenter randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Having sustained a single ischemic or hemorrhagic stroke during the 3- to 12-month period preceding enrollment
* Single stroke
* Inability at the time of screening to demonstrate active extension of the affected metacarpophalangeal and interphalangeal joints at least 10°; and the wrist, 20° (ie, level of impairment that would preclude participation in constraint-induced therapy)
* Score of 47 or lower on the modified 30-item Fugl-Meyer Assessment of UE motor function
* Participants NOT able to extend the affected metacarpophalangeal joints at least 10° and the wrist 20°.

Exclusion Criteria:

* History of carpal tunnel syndrome and conditions that commonly cause peripheral neuropathy, including diabetes, uremia, or associated nutritional deficiencies
* History of head injury with loss of consciousness, severe alcohol or drug abuse, psychiatric illness
* Within 3 months of recruitment, use of drugs known to exert detrimental effects on motor recovery
* Cognitive deficit severe enough to preclude informed consent
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Participants with history of untreated depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Fugl Meyer Assessment | Score change after 18 days of intervention compared to baseline; Score change after 1- and 4-month after the intervention compared to baseline
  The upper extremity FMA is a quantitative measure of motor recovery, sensation, coordination, and speed.

SECONDARY OUTCOMES:
Change in Action Arm Research Test (ARAT) | Score change after 18 days of intervention compared to baseline; Score change after 1- and 4-month after the intervention compared to baseline
  The ARAT was developed specifically to measure UE changes and consists of 4 specific tests to measure grasp, grip, pinch, and gross movement.
Change in Wolf Motor Function Test (WMFT) | Score change after 18 days of intervention compared to baseline; Score change after 1- and 4-month after the intervention compared to baseline
  The WMFT is a time- and function-based evaluation encompassing a battery of 17 tasks
Change in Stroke Impact Scale (SIS) | Score change after 18 days of intervention compared to baseline; Score change after 1- and 4-month after the intervention compared to baseline
  The SIS is a self-report measure that includes 64 items assessing 8 domains including strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrico C, Westgate PM, Salmon Powell E, Chelette KC, Nichols L, Pettigrew LC, Sawaki L. Nerve Stimulation Enhances Task-Oriented Training for Moderate-to-Severe Hemiparesis 3-12 Months After Stroke: A Randomized Trial. Am J Phys Med Rehabil. 2018 Nov;97(11):808-815. doi: 10.1097/PHM.0000000000000971. PMID 29794530